CLINICAL TRIAL: NCT02247336
Title: Impact of Family History and Decision Support on High-risk Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 12-378
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Results first posted 2021-08-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; early detection of cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate (Experimental): Patients will complete a family health history platform at enrollment
  Interventions: Behavioral: Family health history platform (MeTree)
- Delayed (Active Comparator): Patients will complete a family health history platform 12 months following enrollment
  Interventions: Behavioral: Family health history platform (MeTree)

INTERVENTIONS:
Behavioral: Family health history platform (MeTree) — Participants will enter their family health history information into a family health history platform, patients and providers will receive a decision support document and pedigree

SUMMARY:
Family health history can help identify patients at higher than average risk for disease. There is no standardized system for collecting and updating family health history, using this information to determine a patient's disease risk level, and providing screening recommendations to patients and providers. Patients will enter their family health history into MeTree, a family history software program. The program will produce screening recommendations tailored to the patient's family health history. The investigators will examine whether this process increases physician referrals for, and patient uptake of, guideline-recommended screening for colorectal cancer.

DETAILED DESCRIPTION:
Eligible patients are aged 40-65 years, enrolled in primary care, do not have a personal history of colorectal cancer, and have some knowledge of family health history. In Aim 1, a retrospective chart review will be conducted to determine the baseline rate of documenting family health history of colorectal cancer in the medical record for patients enrolled in the Aim 2 randomized trial. In Aim 2, consented patients will be randomized to provide patient-entered family health history and receive patient and provider decision support at enrollment or 12 months later (wait-list control). The primary outcome is risk-appropriate CRC screening/surveillance referral for patients 12 months post-enrollment. Secondary outcomes include patient uptake of recommendations and referral for genetic consultation 12 months post-enrollment. In Aim 3, qualitative interviews will be conducted with physicians and clinic leaders; data will be analyzed using conventional content analysis. In Aim 4, data will be obtained from the administrative databases and patient medical records to conduct a budget impact analysis.

ELIGIBILITY:
Inclusion Criteria:

Primary care provider inclusion criteria:

* primary care physician,
* physician assistant, or nurse practitioner;
* at least one half-day of primary care clinic per week.

Patient inclusion criteria:

* assigned to an enrolled PCP;
* English as preferred language;
* no plans to relocate or leave the VA system in the next 12 months;
* at least one primary care appointment in the 18 months prior to enrollment;
* upcoming PCP appointment with assigned PCP;
* aged 40-64 years; no previous history of colorectal cancer or adenomatous polyps or inflammatory bowel disease;
* no endoscopy within previous 3 years; some knowledge of family health history

Exclusion Criteria:

n/a (contained within inclusion criteria)

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 505 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine I. Voils, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goldstein KM, Fisher DA, Wu RR, Orlando LA, Coffman CJ, Grubber JM, Rakhra-Burris T, Wang V, Scheuner MT, Sperber N, Datta SK, Nelson RE, Strawbridge E, Provenzale D, Hauser ER, Voils CI. An electronic family health history tool to identify and manage patients at increased risk for colorectal cancer: protocol for a randomized controlled trial. Trials. 2019 Oct 7;20(1):576. doi: 10.1186/s13063-019-3659-y. PMID 31590688
- [Derived] Voils CI, Coffman CJ, Wu RR, Grubber JM, Fisher DA, Strawbridge EM, Sperber N, Wang V, Scheuner MT, Provenzale D, Nelson RE, Hauser E, Orlando LA, Goldstein KM. A Cluster Randomized Trial of a Family Health History Platform to Identify and Manage Patients at Increased Risk for Colorectal Cancer. J Gen Intern Med. 2023 May;38(6):1375-1383. doi: 10.1007/s11606-022-07787-9. Epub 2022 Oct 28. PMID 36307642

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate: Patients will complete MeTree at enrollment
  MeTree: Participants will enter their family health history information into MeTree, patients and providers will receive a decision support document and pedigree
- Delayed: Patients will complete MeTree 12 months following enrollment
  MeTree: Participants will enter their family health history information into MeTree, patients and providers will receive a decision support document and pedigree
Period: Overall Study
Arm/Group | Immediate | Delayed
Started | 252 | 253
Completed | 252 | 253
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate | Delayed | Total
Number analyzed (Participants) | 252 | 253 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (7.1) | 51.3 (7.7) | 51.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 28 | 84
  Male | 196 | 225 | 421
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 242 | 240 | 482
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 77 | 87 | 164
  White | 156 | 139 | 295
  More than one race | 9 | 12 | 21
  Unknown or Not Reported | 7 | 9 | 16
Ever had a colonoscopy or sigmoidoscopy [Count of Participants; unit: Participants] | 101 | 97 | 198

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Provider Referral for Risk-appropriate Colorectal Cancer Screening
Description: Patients who receive guideline-recommended referral consistent with the risk stratum determined by the family health history platform.
Time Frame: 12 months
Population: The analysis sample is the number of patients who completed the family health history assessment, as risk level was necessary to determine risk-appropriate referrals.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 252 | 253
Participants | 219 | 232
Statistical Analysis 1: Comparison: Immediate vs Delayed; Using alpha=0.05, 80% power, and a risk-appropriate screening referral rate for the delayed arm ranging from 60% to 70%, n = 250 participants with a completed a family health history assessment per arm with 40 providers was needed to detect differences between arms in appropriate referral ranging from 12% to 13.2%. Sample size calculations accounted for provider clustering using an intra-class correlation coefficient of 0.02 to adjust variance for a Z-test of the difference of two proportions; Test type: Superiority; p = 0.16, Regression, Logistic — A priori threshold was 0.05; generalized estimating equation; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.4 to 1.2] — Generalized estimating equation models were used with a logit link function and an exchangeable correlation structure to account for clustering of participants within provider. Fay and Graubard small sample bias correction was applied

2. Secondary Outcome: Number of Participants Who Received Recommended Colorectal Cancer Screening
Description: Among patients who received a referral, the percentage who received recommended colorectal cancer screening.
Time Frame: 12 months
Population: Analytic sample is participants who had a referral for colorectal cancer screening
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 103 | 109
Participants | 55 | 68
Statistical Analysis 1: Comparison: Immediate vs Delayed; Test type: Superiority; p = 0.23, Regression, Logistic — The a priori threshold was 0.05; generalized estimating equation; Odds Ratio (OR) = 0.7, 95% CI 2-sided [.04 to 1.2] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Patients Who Received Referral for Genetic Consultation
Description: Of patients who received a recommendation for genetic consultation based on the family history platform, the percentage who received a referral for genetic consultation.
Time Frame: 12 months
Population: Subgroup of veterans who received a recommendation for genetic counseling from the family health history platform
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 22 | 15
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Immediate: Patients completed the family history platform at enrollment
  Participants entered their family health history information into the family history platform, and patients and providers received a decision support document and pedigree
- Delayed: Patients completed the family history platform 12 months following enrollment
  Participants entered their family health history information into the family history platform, and patients and providers received a decision support document and pedigree
Arm/Group | Immediate | Delayed
All-Cause Mortality (participants affected / at risk) | 2/252 | 0/253
Serious Adverse Events (participants affected / at risk) | 0/252 | 0/253
Other Adverse Events (participants affected / at risk) | 0/252 | 0/253

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT02247336/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT02247336/ICF_001.pdf